CLINICAL TRIAL: NCT01555996
Title: Early Occupational Therapy (OT) for Delirium Prevention in Older Patients Admitted to Critical Care Unit (CCU)
Brief Title: Early Occupational Therapy for Delirium Prevention in Older Patients Admitted to Critical Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government); National Fund for Research and Development in Health, Chile (Other)
Responsible Party: Principal Investigator, Evelyn Alvarez Espinoza, OT, Principal Investigator, E Alvarez, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SA10I20015
Record Dates: First submitted 2012-01-10; First posted 2012-03-16 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Delirium; Alteration of Cognitive Function; Incompetence, Functional
Keywords: older; delirium; cognitive status; occupational therapy; critically ill patients
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early and intensive OT (Experimental)
  Interventions: Behavioral: Early and Intensive Occupational Therapy
- Standard non-pharmacological prevention (Active Comparator)
  Interventions: Behavioral: Standard non-pharmacological delirium prevention

INTERVENTIONS:
Behavioral: Early and Intensive Occupational Therapy — Intervention group:Standard non-pharmacological prevention plus early and intensive OT. Begin in the first 24 hours in CCU admission. OT areas:1)Multi-sensory stimulation:Intense external stimulation, increase alertness,2)Positioning: Fixtures like dorxi-flexion splints, devices for preventing edema,etc,3)Cognitive Stimulation: Awareness, orientation, attention, memory, calculation, praxis and language,4)Training Activities of Daily Living (ADL): Keep a daily routine and independence in hygiene, grooming and feeding,5)Upper Limb Motor Stimulation (ULMS): Activate functional movement and strength ,6)Family involvement.
  General Guidelines for intervention: Visit of an OT twice a day, 40 minutes each time, for 5 days; meeting of family training for promote strategies during the daily visit.
  Other Names: Active hospital routine
  Arms: Early and intensive OT
Behavioral: Standard non-pharmacological delirium prevention — Non-pharmacological strategies are the first line of approach in the prevention of delirium. It is recommended to implement some of these strategies, which are: Reorientation protocol, including information 4 times a day about time, date, place and reason for hospitalization; early mobilization by physical therapist 3 times a day, corrected sensory impairment (use such as eyeglasses, hearing aids); environment management, use clock and calendar in the patient´s room, promote supervision of a professional or family to avoid physical restraints; sleep protocol, like lower light, noise and nighttime drug administration and finally, reduction of any anticholinergic drugs and minimize the use of benzodiazepines.
  Other Names: Recommended non-pharmacological treatment
  Arms: Standard non-pharmacological prevention

SUMMARY:
This is a randomized, controlled trial to compare the efficacy of two strategies of non-pharmacological prevention of delirium in critically non-ventilated older patients:

* standard non-pharmacological prevention
* intensive nonpharmacological prevention (standard non-pharmacological prevention plus early and intensive occupational therapy).

DETAILED DESCRIPTION:
Delirium is a complication in older, with incidences 70-87% in CCU. This increases mortality, hospital stay, hospital cost, and cognitive impairment. Occupational Therapy (OT) improves independence at discharge, and reduction in delirium in patients undergoing mechanical ventilation. This study compares the efficacy of non pharmacological standard prevention (control group) versus intensive nonpharmacological prevention (experimental group) in the delirium duration in older admitted CCU.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years.
* Admission to CCU for monitoring by acute or chronic illness, expected more than 24 hours
* Informed consent of patient or family related.

Exclusion Criteria:

* Cognitive impairment before to admission (measured by Test Reporter-TIN).
* Severe disorder of communication and cultural constraint of language (inhability of properly communicating in Spanish)
* Delirium at CCU admission or at the beginning of the intervention
* Need for mechanical ventilation
* Early limitation of therapeutic efforts and greater comorbidity with expected mortality within 90 days (in the opinion of the treating team).

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate Delirium duration | From second until sixth days hospitalization
  Twice a day evaluation for delirium with CAM instrument, for 5 days from enrollment

SECONDARY OUTCOMES:
Delirium incidence | From second until sixth days hospitalization
  Proportion of patients in each arm, to developed delirium during daily evaluation
Functional independence | To seventh day of hospitalization and 72 hours before discharge
  Comparing performance of Activity Daily Living (ADL) at hospital discharge compared to baseline, using FIM (Functional Independence Measure) instrument
Strenght of Grip evaluation | To seventh day of hospitalization and 72 hours before discharge
  Strength of grip by Jamar Dynamometer, is evaluated to hospitalary discharge
Cognitive State | To seventh day of hospitalization and 72 hours before discharge
  MMSE (Mini-Mental State Examination), evaluates cognitive state at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Alvarez, Principal Investigator — University of Chile; Maricel Garrido, Study Chair — University of Chile; Eduardo Tobar, Study Chair — University of Chile; Rolando Aranda, Study Chair — University of Chile
Locations (1):
- Hospital Clinico Universidad de Chile, Santiago, RM, Chile